CLINICAL TRIAL: NCT02242552
Title: Personalized Targeted Therapy in Refractory or Relapsed Cancer in Childhood(TRICEPS Study)
Brief Title: Personalized Targeted Therapy in Refractory or Relapsed Cancer in Childhood
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Dr Monia Marzouki, Hematologist/Oncologist, St. Justine's Hospital
Other Study IDs: Triceps
Record Dates: First submitted 2014-08-15; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-08

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, saliva, tumor sample (bone marrow or solid tumors)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A new research paradigm that involves sequencing tumor DNA/RNA to identify driver mutations, select among the Health Canada approved drugs (for adult cancers) known to block certain oncogenic pathways, and recommend these drugs to the treating physician, without taking into account the tumor histology.

In this paradigm, the treatment is targeted to the actionable mutation(s) i.e. those driving oncogenesis. It is also personalized to the molecular signature of the patient's tumor, irrespective of its histopathological subtype. The experience of the investigators team in genomics, including next generation sequencing and bioinformatic analysis combined with the clinical expertise, bring at last this approach within our technical capacities. In parallel, the number of Health Canada-approved drugs (which have been tested in a pediatric setting) designed to interfere with oncogenesis pathways is increasing exponentially.

ELIGIBILITY:
Inclusion Criteria:

At the time of enrollment:

* 21 year-old or less
* Poor prognosis biopsy-proven cancer of any type :
* Cancer (at initial diagnosis) known to be refractory to treatment
* Or cancer refractory to treatment
* Or relapsed cancer
* Written informed consent by patient, parents, or the legal guardians

Exclusion Criteria:

* Estimated life expectancy of less than 3 months.

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents with Relapse or refractory leukemia and solid tumor
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of performing genomic data-based targeted therapy clinical trials in childhood cancers with poor prognosis, including relapsed or refractory cancers. | 24 months
  The study team will evaluate the timeline between decision of biopsy, the actual biopsy, availability of results of the whole-genome analysis, interpretation of results and divulgation of results to patient and family.

SECONDARY OUTCOMES:
Number of children with cancer who are suitable candidates for targeted therapy at our institution each year. | 24 months
Number and type of driver mutation(s) found in our population of recurrent or refractory cancers. | 24 months
Number of cancer patients who harbour actionable driver mutation(s) that can be targeted with a Health Canada approved targeted drug. | 24 months
Feasibility of performing whole genome sequencing and data analysis, identifying a drug based on the genomic data and offering this information to the medical team, the patient and the family within 10-week time frame from diagnosis | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Monia Marzouki, MD, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada